CLINICAL TRIAL: NCT06079463
Title: Determining the Effect of Progressive Relaxation Exercise on Anxiety and Quality of Life in Diabetes Patients
Brief Title: The Effect of Progressive Relaxation Exercise on Anxiety and Quality of Life of Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Gazi Baran CAMCI, Research Assistant, Department of Nursing Principles, Kahramanmaraş İstiklal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KahramanmarasIstiklalU
Record Dates: First submitted 2023-07-05; First posted 2023-10-12 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Patients
Keywords: Anxiety; Diabetes; Exercise; Quality of Life
MeSH Terms: conditions — Anxiety Disorders; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Intervention Model Description: The experimental group consisted of 52 people (the group in which progressive movements exercises were applied) and the control group consisted of 52 people, a total of 104 people. Patients who meet the sample selection criteria are randomized using the Random Integer Generator method from the Random.org organelle Numbers sub-title. In the randomization, the 1-digit experiment will continue to represent the 2-digit control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic patients undergoing progressive relaxation exercise (Experimental): After the purpose of the study was explained and their verbal and written consents were obtained, a questionnaire including the Beck Anxiety Scale, which includes the socio-demographic characteristics, and the World Health Organization Quality of Life Scale, were applied to the patients in the experimental and control groups. will participate in the research, will be asked, and will be filled in face to face by the responsible researcher. After the progressive relaxation exercise training is given to the experimental group patients, the voice recording containing the commands for the application of the progressive relaxation exercise will be sent to the phone of the patient and/or their relatives. Patients in the experimental group spent an average of 25-30 minutes each day for four weeks. Ongoing exercises will be conducted and followed up. At the end of the fourth week, "Beck Anxiety Scale and World Health Organization Quality of Life Scale" will be applied.
  Interventions: Other: progressive relaxation exercise
- Diabetic patients not applied progressive relaxation exercise (No Intervention): After explaining the purpose of the study and obtaining their verbal and written consents, a questionnaire form including the Beck Anxiety Scale and the World Health Organization Quality of Life Scale, in which the socio-demographic characteristics of the experimental and control group patients who will participate in the research, are asked, will be filled in face to face by the principal researcher.Then, a voice recording containing the commands for the application of the progressive relaxation exercise will be sent to the phone of the volunteer patients in this group and/or their relatives, and they will be informed about how to apply it.

INTERVENTIONS:
Other: progressive relaxation exercise — Step 1: Take a comfortable position (sitting or lying down) and wear comfortable, non-tightening clothes.
  Step 2: Try to relax with eyes closed, without focusing on thoughts, by focusing on your own body muscles.
  Step 3: Right and left, respectively, hands, arms (triceps muscle), chest, abdomen, hips, legs (thigh muscles), feet and toes, neck, shoulder (scapula muscles) and muscle groups on the face (around the eyes, chin) and eyebrow muscles) by concentrating on contracting and relaxing these muscles.
  Step 4: Focusing on the muscle groups of the whole body, contracting and relaxing.
  Step 5: Opening the eyes slowly, trying to feel the feeling of comfort in the body (Turkish Psychologists Association Progressive Relaxation Exercises).
  Arms: Diabetic patients undergoing progressive relaxation exercise

SUMMARY:
Purpose of the study: The study aimed to direct the anxiety and quality of life of progressive movement exercise in diabetic patients.

Type of research: A randomized controlled pre-test-post-test study was planned with the aim of directing progressive movement exercise on anxiety and quality of life in diabetics.

research questions Q1: Does progressive movement exercise have an effect on diabetic anxiety and quality of life? Population of the Research and Sample Selection: The home of the research will be the diabetes windows to the internal service on data collection. G-power 3.1 analysis program environment to calculate large sample size. Sampling of the research; With 0.61% effect sizes, 0.05% error level, 95% confidence interval and 80% power to show the universe, 52 people took part in the experimental motivations (phased training exercises group) and 52 people took part in the control slots, for a total of 104 people. Sample selection criteria patients are randomized using the Random Integer Generator method from the Numbers subheading on the Random.org website. In randomization, aspects will be collected representatively of 1 experimental group and 2 control groups.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is an important health problem all over the world, which mostly starts in middle and advanced ages and has an important place among non-communicable chronic diseases due to its high morbidity and mortality. It can affect the patient biologically, psychologically, socially and psychosexually. In addition, generalized anxiety disorder was observed in 14% of the patients and an increase in anxiety levels was observed in 40%. Meta-analyses have shown that the presence of diabetes in an individual has a 24% risk of developing depression. This increase in depression and anxiety in DM negatively affects the patient's compliance and response to treatment and the prognosis of the disease. In addition, it causes deterioration in self-care and quality of life, the risk of developing complications, morbidity, mortality and health expenditures. Progressive relaxation exercise (PGE) is the voluntary contraction and relaxation of large muscle groups in the body, and noticing the difference. The PGE technique, developed by Jacobson in 1934, is based on the idea that anxiety-provoking thoughts and events create physiological tension. Doctor Edmund Jacobson developed the PGE to raise awareness of skeletal muscle tension. Muscle tension is triggered by various negative emotions and psychosomatic diseases. With this exercise, relaxation is aimed to reduce the feeling of tension and the perceived stress level. Progressive relaxation exercises are an inexpensive method that can be easily taught by nurses, yoga instructors, clinical psychologists, and other complementary alternative medicine practitioners. PGE is performed one-on-one or as a group, in one or several sessions, with the help of a CD or sound recorder. In order to increase its effectiveness, it can be applied with musical accompaniment, visual imagery or diaphragmatic breathing. Deep relaxation can be used to prevent the tensions experienced after stressful events from harming the body; It is one of the physiological and psychological relaxation methods such as sports and sleep. It is very useful for maintaining physical and mental health. It is suggested that a deep relaxation exercise that usually lasts 25-30 minutes can provide a benefit close to the benefit of two hours of deep sleep. In the literature, it is stated that if these exercises can be performed consistently and systematically for a long time, they have positive effects on stress-based insomnia, migraine pain, diabetes and high blood pressure. When we look at the literature, it has been determined that progressive relaxation exercises have a positive effect on anxiety and quality of life in many disease groups, but it has been observed that there are not enough studies in which these exercises are applied in diabetes patients and their effects on anxiety and quality of life are examined. The research is important in that it will examine the effect of progressive relaxation exercises on anxiety and quality of life, which is essential for diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients who will be treated in the Internal Medicine Service who want to participate in the study voluntarily.
* Patients over the age of 18

Exclusion Criteria:

* Patients who do not want to participate in the study.
* Patients who are unable to perform the progressive relaxation exercise (amputation, etc.).
* Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Scale | 4 weeks
  Progressive relaxation exercise was applied to the patients for 4 weeks. After the application, anxiety scores were determined with the Back Anxiety Scale and the results were recorded.

SECONDARY OUTCOMES:
World Health Organization Quality of Life Scale | 4 weeks
  Progressive relaxation exercise was applied to the patients for 4 weeks. After the application, quality of life scores were determined with the World Health Organization Quality of Life Scale and the results were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Üniversitesi, Erzurum, Turkey (Türkiye)